CLINICAL TRIAL: NCT00977340
Title: Psychotherapeutic Treatment of Chronic Nightmares: Differential Efficacy of Imagery Rehearsal Therapy Compared to Confrontation and Psychotherapeutic Placebo
Brief Title: Study on the Psychotherapeutic Treatment of Chronic Nightmares
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Regina Steil, Scientific director behavior therapy outpatient center, Goethe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: StudieAlptraum1
Record Dates: First submitted 2009-09-14; First posted 2009-09-15 (Estimated); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Nightmare Disorder
Keywords: Chronic nightmare sufferers; nightmares; Imagery Rehearsal Therapy IRT; sleep disturbance; treatment of nightmares; confrontation; People who suffer of chronic nightmares
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Imagery Rehearsal Treatment (Experimental): Imagery Rehearsal Treatment; 1 session on-site and 4 weeks of individual daily training; following principles Krakow and Zadra (2006)
  Interventions: Behavioral: Imagery Rehearsal Treatment
- Confrontation (Experimental): Confrontation with nightmare content, until fear reaction habituates; 1 session on-site and 4 weeks of individual daily training
  Interventions: Behavioral: confrontation
- Imagination (Placebo Comparator): Imagination of a safe and pleasant site; 1 session on-site and 4 weeks of individual daily training
  Interventions: Behavioral: imagination

INTERVENTIONS:
Behavioral: Imagery Rehearsal Treatment — Imagery Rehearsal Therapy
  Arms: Imagery Rehearsal Treatment
Behavioral: confrontation — Confrontation
  Arms: Confrontation
Behavioral: imagination — Imagination
  Arms: Imagination

SUMMARY:
The purpose of this study is to determine whether a change in the content of nightmares is necessary at all in the treatment of chronic nightmares or if a single confrontation with their content is sufficient to reduce nightmare frequency significantly.

DETAILED DESCRIPTION:
The inclusion and exclusion criteria are assessed during a telephone interview. If the participants meet the criteria, they are randomly assigned to two intervention groups or an active control group. In the first session the participants who suffer from chronic nightmares are interviewed using the Structured Clinical Interview for DSM-IV (SCID-I and -II) to determine the clinical diagnosis; in addition, they are given questionnaires and record sheets to obtain baseline data. They are asked to record their nightmares in a "dream diary" up until the next session four weeks later. At that session they learn one of three interventions to reduce nightmares. The first group receives imagery rehearsal treatment in which participants learn to consciously alter the contents of their nightmares and then to visualize the new set of images. The second group is subjected to confrontation treatment in which they are instructed to confront their nightmares until habituation. The third group, the psychotherapeutic placebo group, just learn an imagination technique, without reference to their nightmares. At the end of the intervention session all participants receive written instructions on how to perform the learned method at home. They must also record their dreams up until the next session. That session and the last one are used for data acquisition. At these sessions, the participants are asked to fill in the questionnaires given to them at the beginning of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* nightmare frequency of at least one night per week for six month duration
* stable medication
* if currently in psychotherapy: no treatment of nightmares
* Informed consent

Exclusion Criteria:

* Life time clinical diagnosis of schizophrenia, schizoaffective disorder or bipolar disorder according to DSM-IV
* Body mass index < 17
* Initiation of nightmares after taking pharmaceuticals
* Clinical diagnosis of alcohol or drug addiction according to DSM-IV
* Mental retardation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2017-11-08 (Actual); Study Completion 2017-11-08 (Actual)

PRIMARY OUTCOMES:
frequency of nightmares | in the first diagnostical session, four weeks after interventional session in addition to follow-up-measurement
  Nightmare Frequency Questionnaire (NFQ, Krakow et al., 2000) number of nightmares per week. The participant is asked to state the number of nightmares in the last three months, the response is to be given as an absolute frequency per year, month, or week, whichever is applicable. The range is zero to any number the participant states, the maximum number reported was 20.
nightmare effects | in the first diagnostical session, four weeks after interventional session in addition to follow-up-measurement
  Nightmare Effects Survey (NES, Krakow et al., 2000) The first item asks whether the person's life is generally affected by nightmares. The remaining eleven items list areas in daily life (sleep, work, relationships, daytime energy, school, mood, sex life, diet, mental health, physical health, and leisure activities) rated on 5-point Likert scales regarding how much they are "adversely or negatively affected by nightmares". The range is 0 to 44, and higher values indicate more effects.
nightmare distress | in the first diagnostical session, four weeks after interventional session in addition to follow-up-measurement
  Nightmare Distress Questionnaire (NDQ, Belicki, 1992) The NDQ consists of 13 items rated on 5-point Likert scales. Eleven items pertain to daytime consequences of nightmares (e.g., disliking someone because they were in a nightmare; being afraid to fall asleep for fear of having a nightmare); two items explore interest in professional help and treatment. The range is 13 to 65, and higher values indicate more distress.

SECONDARY OUTCOMES:
Anxiety | in the first diagnostical session, four weeks after interventional session in addition to follow-up-measurement
  self rated: Beck Anxiety Inventory: 21 Items to be rated on 0 to 3 scales, range 0 to 63, higher values indicate higher anxiety in both measures rated by therapist on Hamilton Anxiety Scale: 14 Items to be rated on 5-point-scales from "not at all" to "very strong", range 0 to 56
Depression | in the first diagnostical session, four weeks after interventional session in addition to follow-up-measurement
  self rated: Beck Depression Inventory II, 21 Items to be rated on 0 to 3 scales, range 0 to 63 rated by therapist on Hamilton Depression Scale, 21 Items to be rated on 0-2 or 0-4 scales, range 0-66, higher values indicate higher depression in both measures
sleep quality | in the first diagnostical session, four weeks after interventional session in addition to follow-up-measurement
  Landeck Inventory for the Assessment of Sleep Disorders (LISST, Weeß, 2002): This is a screening instrument for sleep disorders, only the item measuring dream recall and the 8-item sleep quality subscale were used. Both use 6-point Likert scales. The sleep quality subscale score range is 0 to 40, and higher values indicate lower sleep quality.
self efficacy | in the first diagnostical session, four weeks after interventional session in addition to follow-up-measurement
  Selbstwirksamkeitsskala (General self efficacy, Jerusalem & Schwarzer, 1998) This 10-item measure contains statements such as "I am confident that I could deal efficiently with unexpected events" or "I can usually handle whatever comes my way" rated on 4-point Likert scales. The scale was used to operationalize mastery. Its range is 10 to 40, with higher values indicating higher self-efficacy.
General psychopathology | in the first diagnostical session, four weeks after interventional session in addition to follow-up-measurement
  Symptom Checklist 90-R The SCL measures a wide variety of psychopathological symptoms. The Global Severity Index (GSI) was used. Its range is 0 to 4, with higher values indicating more and/or more intense symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Regina Steil, PhD, Principal Investigator — Johann Wolfgang Goethe University - Department of Clinical Psychology and Ppsychotherapy
Locations (1):
- Johann Wolfgang Goethe University - Department of Clinical Psychology and Ppsychotherapy, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No